CLINICAL TRIAL: NCT02008279
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Pharmacokinetics and Safety of CNTO3157 Following an Escalating Single SC Dose to Healthy Japanese and Caucasian Subjects or a Single Intravenous Dose to Healthy Caucasian Subjects
Brief Title: A Safety and Pharmacokinetics Study of CNTO 3157 in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102823; CNTO3175NAP1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy; CNTO 3157; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group 1A (Experimental): 100 mg CNTO 3157 or placebo in healthy male Japanese participants
  Interventions: Biological: 100 mg CNTO 3157; Drug: Placebo
- Group 1B (Experimental): 100 mg CNTO 3157 or placebo in healthy male Caucasian participants
  Interventions: Biological: 100 mg CNTO 3157; Drug: Placebo
- Group 2A (Experimental): 300 mg CNTO 3157 or placebo in healthy male Japanese participants
  Interventions: Biological: 300 mg CNTO 3157; Drug: Placebo
- Group 2B (Experimental): 300 mg CNTO 3157 or placebo in healthy male Caucasian participants
  Interventions: Biological: 300 mg CNTO 3157; Drug: Placebo
- Group 3A (Experimental): 600 mg CNTO 3157 or placebo in healthy male Japanese participants
  Interventions: Biological: 600 mg CNTO 3157; Drug: Placebo
- Group 3B (Experimental): 600 mg CNTO 3157 or placebo in healthy male Caucasian participants
  Interventions: Biological: 600 mg CNTO 3157; Drug: Placebo
- Group 4 (Experimental): 300 mg CNTO 3157 in healthy male Caucasian participants
  Interventions: Biological: 300 mg CNTO 3157

INTERVENTIONS:
Biological: 100 mg CNTO 3157 — A single subcutaneous (SC) (under the skin) injection of 100 mg CNTO 3157
  Arms: Group 1A; Group 1B
Biological: 300 mg CNTO 3157 — 2 SC injections of CNTO 3157 providing a total dose of 300 mg
  Arms: Group 2A; Group 2B
Biological: 600 mg CNTO 3157 — 4 SC injections of CNTO 3157 providing a total dose of 600 mg
  Arms: Group 3A; Group 3B
Biological: 300 mg CNTO 3157 — 300 mg of CNTO 3157 as an intravenous (IV) infusion (into a vein) administered over a period of 30 minutes
  Arms: Group 4
Drug: Placebo — SC injections of placebo (number of injections to equal number of injections of CNTO 3157)
  Arms: Group 1A; Group 1B; Group 2A; Group 2B; Group 3A; Group 3B

SUMMARY:
The purpose of this study is to find out if different doses of CNTO 3157 are well tolerated in both Japanese and Caucasian men as well as to understand how the body absorbs and removes the study drug after being injected or infused into the body.

DETAILED DESCRIPTION:
This will be a randomized (the treatment is assigned by chance), double-blind (neither the participants nor study staff know the identity of the assigned treatment), placebo-controlled study (one of the study medications is inactive) to investigate the pharmacokinetics (ie, how the body absorbs and removes the study drug) and safety of subcutaneous (administered under the skin) (SC) CNTO 3157 (a drug currently being investigated for the treatment of asthma) in both Japanese and Caucasian men. Additionally, an open-label cohort (where participants and study staff know the identity of the assigned treatment) in Caucasian men will investigate the pharmacokinetics and safety of a single intravenous (into a vein) (IV) infusion. The study will consist of 3 phases: a screening phase, a treatment phase (comprising 2 days and 1 night at the study center) and a follow-up period (comprising approximately 11 visits to the study center). During the double-blind SC treatment period, participants will be randomly assigned to 1 of 3 treatment groups: group 1 will receive a single SC injection of 100 mg CNTO 3157 or placebo; group 2 will receive 2 SC injections of CNTO 3157 (making a total dose of 300mg) or placebo; group 3 will receive 4 SC injections of CNTO 3157 (making a total dose of 600 mg) or placebo. Group 4 (open-label cohort) will receive a single IV infusion of 300 mg CNTO 3157. Participants will be enrolled in each SC dose group sequentially from the lower to higher dose level. The study sponsor and the study doctor will review the test results (in terms of safety and tolerability) for each group before dosing participants in the next treatment group; this review will be carried out in a blinded manner. An equal number of Japanese and Caucasian participants will be assigned to the SC treatment groups forming 2 subgroups within each group (groups 1A, 1B, 2A, 2B, 3A and 3B). Within each SC treatment group, 10 participants will be randomly assigned in a 4 to 1 ratio to receive CNTO 3157 or placebo. Only Caucasian participants will be enrolled in the IV treatment group (group 4). For each treatment group, blood and urine samples will be taken at various time points during the study. Each participant will take part in the study for approximately 85 days. Participant safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a screening body weight in the range of 50 kg to 100 kg, inclusive, and a screening body mass index of 18.5 kg/m2 to 30 kg/m2, inclusive
* Participants must be: of Japanese descent whose parents and maternal and paternal grandparents are Japanese, as determined by participant's verbal report; Japanese participants must have valid government issued identification; Japanese participants must have resided outside of Japan for <= 5 years; or must be of non-Hispanic Caucasian descent whose parents are Caucasian, as determined by participant's verbal report
* Participants must have been exposed to herpes simplex-type 1 virus (HSV-1) as documented by a positive serology test result for HSV-1 performed at screening, but have no signs or symptoms suggestive of an active HSV-1 infection and are not receiving prescription treatment or prophylaxis for HSV-1

Exclusion Criteria:

* Participant has or has had a clinically significant (viral, bacterial or parasitic) infection, a prior history of recurrent serious infection (eg, sepsis, pneumonia or pyelonephritis) or be immunosuppressed or have been hospitalized or received IV antibiotics for an infection during the 2 months prior to screening
* Participant is infected with human immunodeficiency virus or tests positive for hepatitis B virus infection or has antibodies to hepatitis C virus at screening
* Participant has received any live or attenuated virus or bacterial vaccinations within 3 months prior to study agent administration or is expected to receive any live virus or bacterial vaccinations during the study or up to 6 months after administration of the study agent
* Participant has had major surgery, (eg, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study OR has had a major illness or hospitalization within 1 month prior to study agent administration
* Participant has a history of, or currently active illness/disorder, considered to be clinically significant by the Investigator or any other illness/disorder that the Investigator considers should exclude the participant from the study or that could interfere with the interpretation of the study results

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | Up to Day 57
  The frequency of adverse events will be used to assess the safety and tolerability of CNTO 3157.
Serum concentrations of CNTO 3157 in Caucasian and Japanese participants following single subcutaneous doses of 100 mg, 300 mg, and 600 mg | Up to Day 57
  Serum concentrations of CNTO 3157 will be used to determine pharmacokinetic parameters (measurements that explore what the body does to the drug).
Titer (concentration) of antibodies to CNTO 3157 in Caucasian and Japanese participants following single subcutaneous doses of 100 mg, 300 mg, and 600 mg | Up to Day 57
  Serum samples will be screened for antibodies binding to CNTO 3157 providing an indication of the ability of CNTO 3157 to cause an immune response.

SECONDARY OUTCOMES:
Serum concentrations of CNTO 3157 in Caucasian participants following a single intravenous infusion of 300 mg | Up to Day 57
  Serum concentrations of CNTO 3157 will be used to determine pharmacokinetic parameters (measurements that explore what the body does to the drug).
Titer (concentration) of antibodies to CNTO 3157 in Caucasian participants following a single intravenous infusion of 300 mg | Up to Day 57
  Serum samples will be screened for antibodies binding to CNTO 3157 providing an indication of the ability of CNTO 3157 to cause an immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States